CLINICAL TRIAL: NCT00234663
Title: A Phase 2 Study of PTC124 as an Oral Treatment for Nonsense-Mutation-Mediated Cystic Fibrosis
Brief Title: PTC124 for Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: Cystic Fibrosis Foundation (Other); FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-003-CF; 1R01FD003009-01 (FDA)
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Nonsense mutation; Premature stop codon
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

INTERVENTIONS:
Drug: PTC124

SUMMARY:
In some patients with cystic fibrosis (CF), the disease is caused by a nonsense mutation (premature stop codon) in the gene that makes the cystic fibrosis transmembrane regulator (CFTR) protein. PTC124 has been shown to partially restore CFTR production in animals with CF due to a nonsense mutation. The main purpose of this study is to understand whether PTC124 can safely increase functional CFTR protein in the cells of patients with CF due to a nonsense mutation.

DETAILED DESCRIPTION:
In this study, patients with CF due to a nonsense mutation will be treated with a new investigational drug called PTC124. Evaluation procedures (history, physical examination, blood and urine tests to assess organ function, electrocardiogram (ECG), chest x-ray, and CF-specific tests) to determine if a patient qualifies for the study will be performed within 21 days prior to the start of treatment. Eligible patients who elect to enroll in the study will then participate in two 28-day treatment and follow-up periods (56 days total). Within the first 28-day period, PTC124 treatment will be taken 3 times per day with meals for 14 days at doses of 4 mg/kg (breakfast), 4 mg/kg (lunch) and 8 mg/kg (dinner); there will then be an interval of 14 days without treatment. Within the second 28-day period, PTC124 treatment will be taken 3 times per day with meals for 14 days at doses of 10 mg/kg (breakfast), 10 mg/kg (lunch) and 20 mg/kg (dinner); there will then be an interval of 14 days without treatment. There will be a 2-night stay at the clinical research center at the beginning and at the end of each 14 days of PTC124 treatment, which means that there will be four 2-night stays at the clinical research center during the study. During the study, PTC124 efficacy, safety, and pharmacokinetics will be evaluated periodically with measurement of transepithelial potential difference (TEPD), nasal mucosal brushing to assess for cellular CFTR mRNA and protein, medical history, physical examinations, blood tests, urinalysis, ECGs, chest x-ray, and pulmonary function tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on documented evidence of a conclusively abnormal sweat test (sweat chloride >60 mEq/liter).
* Abnormal chloride secretion as measured by TEPD (a less than -5 mV TEPD assessment of chloride secretion with chloride-free amiloride and isoproterenol).
* Presence of a nonsense mutation in one of the alleles of the CFTR gene.
* Age ≥18 years.
* Body weight ≥40 kg.
* FEV1 ≥40% of predicted for age, gender, and height (Knudson standards).
* Oxygen saturation (as measured by pulse oximetry) ≥92% on room air.
* Willingness of male and female patients, if not surgically sterile, to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and follow-up periods.
* Negative pregnancy test (for females of childbearing potential).
* Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, and study restrictions.
* Ability to provide written informed consent.

Exclusion Criteria:

* Prior or ongoing medical condition, medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the patient, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
* Ongoing acute illness including acute upper or lower respiratory infections within 2 weeks before start of study treatment.
* History of major complications of lung disease within 2 months prior to start of study treatment.
* Abnormalities on screening chest x-ray suggesting clinically significant active pulmonary disease other than CF, or new, significant abnormalities that may be indicative of clinically significant active pulmonary involvement secondary to CF.
* Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test.
* Hemoglobin <10 g/dL.
* Serum albumin <2.5 g/dL.
* Abnormal liver function (serum ALT, AST, GGT, alkaline phosphatase, LDH, or total bilirubin > upper limit of normal).
* Abnormal renal function (serum creatinine >1.5 times upper limit of normal).
* Pregnancy or breast-feeding.
* History of solid organ or hematological transplantation.
* Exposure to another investigational drug within 14 days prior to start of study treatment.
* Ongoing participation in any other therapeutic clinical trial.
* Ongoing use of thiazolidinedione peroxisome proliferator-activated receptor gamma (PPAR γ) agonists, eg, rosiglitazone (Avandia® or equivalent) or pioglitazone (Actos® or equivalent)
* Change in intranasal medications (including use of corticosteroids, cromolyn, ipratropium bromide, phenylephrine, or oxymetazoline) within 14 days prior to start of study treatment.
* Change in treatment with systemic or inhaled corticosteroids within 14 days prior to start of study treatment.
* Use or requirement for inhaled gentamicin or amikacin within 14 days prior to start of study treatment or during study treatment.
* Requirement for systemic aminoglycoside antibiotics within 14 days prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
CFTR activity as assessed by nasal transepithelial potential difference (TEPD)

SECONDARY OUTCOMES:
Side effects
Presence of CFTR protein and mRNA
Compliance with treatment
Lung function
PTC124 pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: John P Clancy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - The Children's Hospital, Denver, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio